CLINICAL TRIAL: NCT03780998
Title: Effects of Sodium Pentaborat Based Gel on Perianal Benign Diseases. Prospective Clinical Trial
Brief Title: Effects of Sodium Pentaborat Based Gel on Perianal Benign Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Collaborators: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Erhan Aysan, MD Prof, Yeditepe University
Other Study IDs: yeditepe university
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Hemorrhoids; Anal Fissure; Perianal Fistula
MeSH Terms: conditions — Hemorrhoids; Fissure in Ano

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — histopathological evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group-1 (n: 50): Healthy cases: Control group
  Interventions: Drug: Life7
- Group-2 (n:50): Grade 1 hemorroid: With perianal examination diagnosed of grade 1 hemorroidal disease
  Interventions: Drug: Life7
- Group-3 (n:50): Grade 2 hemorroid: With perianal examination diagnosed of grade 2 hemorroidal disease
  Interventions: Drug: Life7
- Group-4 (n:50): Anal fissure cases: With perianal examination diagnosed of anal fissure cases
  Interventions: Drug: Life7
- Group-5 (n:50): Simple perianal fistula: With perianal examination diagnosed of uncomplicated, simple perianal fistula cases
  Interventions: Drug: Life7

INTERVENTIONS:
Drug: Life7 — Life7 will used on the perianal skin with finger tips
  Other Names: Life 7

SUMMARY:
New produced and patented sodium pantaborat based gel will be use for treatment of benign perianal diseases (hemooroidal disease, anal fissura anda perianal fistula)

DETAILED DESCRIPTION:
Prospective randomised clinical trial planned. Older than 18 years old perianal benign diseases (grade 1 and 2 hemorroidal disease, anal fissura, uncomplicated simple perianal fistula) cases without malign tumour, cronic colorectal disases, and routine used of vasoactive medication cases were entered the study. Younger than 18 years old, diagnosed any malign tumor and/or cronic colorectal disaeses, routine used of vasoact,ve mediaction cases were exclused of the study.

Group-1 (n: 50): Healthy cases (control group) Group-2 (n:50): Grade 1 hemorroidal disease cases Group-3 (n:50): Grade 2 hemorroidal disease cases Group-4 (n:50): Anal fissure cases Group-5 (n:50): Uncomplicated, simple perianal fistula cases

ELIGIBILITY:
Inclusion Criteria:

* Grade 1 and 2 hemorroidal disease
* Cronic anal fissura
* Uncomplicated simple perianal fistula

Exclusion Criteria:

* Any malign tumour
* Cronic colorectal disases
* Routine used of vasoactive medication

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Older than 18 years old cases
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain symtom differences | six months
  Pain Scale from level 1 to level 10.
Lowering of the grade of the hemorroidal disease (hemoroidal disease is four grades; grade 1, grade 2, grade 3, and grade 4) | six months
  Surgeon general physical examination
Closing of anal fissur line | six months
  Surgeon general physical examination. Fissur line is exist or not exist
Lowering of leakage amount of perianal fistule | six months
  Three grade: lower, same, more